CLINICAL TRIAL: NCT05727488
Title: Investigating the Effects of SARAH Exercise Program on Proprioception and Hand Functions in Patients With Rheumatoid Arthritis
Brief Title: SARAH Exercise Program in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Deniz Bayraktar, Assistant Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SARAHRA
Record Dates: First submitted 2023-01-27; First posted 2023-02-14 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Hand; Proprioception; Exercise
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The SARAH exercise program will be delivered by sending messages and video instructions via a freeware and cross-platform messaging service (WhatsApp Messenger) on a weekly basis.
  Interventions: Other: Exercise
- Control (No Intervention): Patients in the control group will not receive any exercise intervention. They will only maintain their routine medical treatment.

INTERVENTIONS:
Other: Exercise — Participants will be asked to practice home exercises every day of the week for 12 weeks. The SARAH exercise program consists of 7 mobility and 4 strengthening exercises. Progress will be made by increasing the repetitions and duration of the exercises every week.
  Arms: Exercise

SUMMARY:
The aim of this study is to investigate the effectiveness of the SARAH home exercise program to be applied for 12 weeks on wrist proprioception and hand functions in adult patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Finger/hand/wrist joints can be affected in the early period in patients with RA, and as the disease progresses, it can significantly limit the patient's functionality. Damage to articular and periarticular structures seen in inflammatory arthritis may affect the sense of proprioception by destroying mechanoreceptors located in these areas. Hand functions may worsen as a result of the worsening of the sense of proprioception, which can be defined as being aware of body parts.

SARAH (Strengthening and Stretching for Rheumatoid Arthritis of the Hand) home exercise program, which is a widely preferred approach in the case of hand involvement in patients with rheumatoid arthritis (RA), includes exercises to increase hand-wrist strength and mobility. Although the effectiveness of this program on pain, muscle strength, and range of motion has been demonstrated in large patient groups, its effect on proprioception and hand functions, which may be caused by inflammatory arthritis, has not been studied. Therefore, this study aims to investigate the effectiveness of the SARAH home exercise program on wrist proprioception and hand functions in adult patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. RA diagnosis according to 2010 ACR/EULAR RA criteria
2. Being between the ages of 18-65
3. Being able to follow Turkish instructions
4. Volunteering to participate in the study

Exclusion Criteria:

1. Being in an acute disease exacerbation period
2. Ongoing physiotherapy/occupational/exercise treatment regarding hands within the last 6 months
3. History of steroid injection, surgery, or trauma to the upper extremity in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Change in Wrist Joint Position Sense | At baseline and twelve weeks later
  Wrist joint position sense will be evaluated with joint position sense goniometry. Joint position sense is measured by the ability to actively repeat a predetermined target angle. During the measurement, the wrist of the participant will passively be brought to the target angle and be kept in this position for three seconds. The participant will be asked to keep this position in his/her memory, then the wrist will passively be brought to the starting position. Then, the participant will be requested to bring her/his hand actively to these predetermined position. Wrist movements will be determined as three repetitive measurements for flexion, extension, radial deviation, and ulnar deviation directions.
Change in Hand Performance | At baseline and twelve weeks later
  Hand performance will be evaluated Nine-Hole Peg Test.
Change in Grip Strength | At baseline and twelve weeks later
  Hand grip strength will be evaluated with a hand-dynamometer.
Change in Pinch Strength | At baseline and twelve weeks later
  Pinch strength will be evaluated by using a pinchmeter.
Change in Self-reported Hand Functions | At baseline and twelve weeks later
  Duruoz Hand Index and The Measures of Activity Performance of the Hand Questionnaire will be used for subjective assessment of hand functions. Higher scores in both questionnaires reflect poorer hand functions.

SECONDARY OUTCOMES:
Change in Pain | At baseline and twelve weeks later
  Numeric rating scale (NRS) will be used for pain assessment. NRS is scored between 0-10 and, higher scores indicate higher level of pain.
Change in Morning Stiffness | At baseline and twelve weeks later
  Morning stiffness related to the hand/wrist of the patients will be questioned by using Numeric Rating Scale (0-10) in terms of duration and severity. Higher scores indicate worse morning stiffness.
Change in Disease Activity | At baseline and twelve weeks later
  Disease Activity 28 C-Reactive Protein (DAS28-CRP) will be used to evaluate disease activity.
Change in General Functioning | At baseline and twelve weeks later
  Health Assessments Questionnaire-Disability Index, which is a self-report tool and has 20 items, will be used to evaluate the general functioning. All items are scored between 0 and 3. All scores are summed and divided by 20 to obtain a total score (0-3). Higher scores indicate a worse functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Bayraktar, PT, PhD, Principal Investigator — Izmir Katip Celebi University
Locations (1):
- Izmir Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable requests.
Time Frame: Data will be available after completing the study and will be available for 20 years.
Access Criteria: Data will be shared for only academic purposes (for conducting a meta-analysis or a systematic review)

REFERENCES:
- [Background] Figus FA, Piga M, Azzolin I, McConnell R, Iagnocco A. Rheumatoid arthritis: Extra-articular manifestations and comorbidities. Autoimmun Rev. 2021 Apr;20(4):102776. doi: 10.1016/j.autrev.2021.102776. Epub 2021 Feb 17. PMID 33609792
- [Background] Kopruluoglu M, Naz I, Solmaz D, Akar S. Hand functions and joint position sense in patients with psoriatic arthritis- a comparison with rheumatoid arthritis and healthy controls. Clin Biomech (Bristol). 2022 May;95:105640. doi: 10.1016/j.clinbiomech.2022.105640. Epub 2022 Apr 4. PMID 35405540
- [Background] Bearne LM, Coomer AF, Hurley MV. Upper limb sensorimotor function and functional performance in patients with rheumatoid arthritis. Disabil Rehabil. 2007 Jul 15;29(13):1035-9. doi: 10.1080/09638280600929128. PMID 17612988
- [Background] Smolen JS, Aletaha D, McInnes IB. Rheumatoid arthritis. Lancet. 2016 Oct 22;388(10055):2023-2038. doi: 10.1016/S0140-6736(16)30173-8. Epub 2016 May 3. PMID 27156434
- [Background] Williams MA, Srikesavan C, Heine PJ, Bruce J, Brosseau L, Hoxey-Thomas N, Lamb SE. Exercise for rheumatoid arthritis of the hand. Cochrane Database Syst Rev. 2018 Jul 31;7(7):CD003832. doi: 10.1002/14651858.CD003832.pub3. PMID 30063798
- [Background] Heine PJ, Williams MA, Williamson E, Bridle C, Adams J, O'Brien A, Evans D, Lamb SE; SARAH Team. Development and delivery of an exercise intervention for rheumatoid arthritis: strengthening and stretching for rheumatoid arthritis of the hand (SARAH) trial. Physiotherapy. 2012 Jun;98(2):121-30. doi: 10.1016/j.physio.2011.03.001. PMID 22507362
- [Background] Lamb SE, Williamson EM, Heine PJ, Adams J, Dosanjh S, Dritsaki M, Glover MJ, Lord J, McConkey C, Nichols V, Rahman A, Underwood M, Williams MA; Strengthening and Stretching for Rheumatoid Arthritis of the Hand Trial (SARAH) Trial Team. Exercises to improve function of the rheumatoid hand (SARAH): a randomised controlled trial. Lancet. 2015 Jan 31;385(9966):421-9. doi: 10.1016/S0140-6736(14)60998-3. Epub 2014 Oct 9. PMID 25308290
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Background] Jensen Hansen IM, Asmussen Andreasen R, van Bui Hansen MN, Emamifar A. The Reliability of Disease Activity Score in 28 Joints-C-Reactive Protein Might Be Overestimated in a Subgroup of Rheumatoid Arthritis Patients, When the Score Is Solely Based on Subjective Parameters: A Cross-sectional, Exploratory Study. J Clin Rheumatol. 2017 Mar;23(2):102-106. doi: 10.1097/RHU.0000000000000469. PMID 27870649
- [Background] Duruoz MT, Poiraudeau S, Fermanian J, Menkes CJ, Amor B, Dougados M, Revel M. Development and validation of a rheumatoid hand functional disability scale that assesses functional handicap. J Rheumatol. 1996 Jul;23(7):1167-72. PMID 8823687
- [Background] Earhart GM, Cavanaugh JT, Ellis T, Ford MP, Foreman KB, Dibble L. The 9-hole PEG test of upper extremity function: average values, test-retest reliability, and factors contributing to performance in people with Parkinson disease. J Neurol Phys Ther. 2011 Dec;35(4):157-63. doi: 10.1097/NPT.0b013e318235da08. PMID 22020457
- [Background] Hamilton GF, McDonald C, Chenier TC. Measurement of grip strength: validity and reliability of the sphygmomanometer and jamar grip dynamometer. J Orthop Sports Phys Ther. 1992;16(5):215-9. doi: 10.2519/jospt.1992.16.5.215. PMID 18796752
- [Background] Haidar SG, Kumar D, Bassi RS, Deshmukh SC. Average versus maximum grip strength: which is more consistent? J Hand Surg Br. 2004 Feb;29(1):82-4. doi: 10.1016/j.jhsb.2003.09.012. PMID 14734079
- [Background] Halpern CA, Fernandez JE. The effect of wrist and arm postures on peak pinch strength. J Hum Ergol (Tokyo). 1996 Dec;25(2):115-30. PMID 9735592
- [Background] Leung YY, Tillett W, Hojgaard P, Orbai AM, Holland R, Mathew AJ, Goel N, Chau J, Lindsay CA, Ogdie A, Coates LC, Christensen R, Mease PJ, Strand V, Gladman DD. Test-retest Reliability for HAQ-DI and SF-36 PF for the Measurement of Physical Function in Psoriatic Arthritis. J Rheumatol. 2021 Oct;48(10):1547-1551. doi: 10.3899/jrheum.210175. Epub 2021 Apr 15. PMID 33858982